CLINICAL TRIAL: NCT03666754
Title: The Effectiveness of Compression and Early Glue Ablation of Saphenous Vein Reflux Compared With Compression Alone in the Healing of Venous Ulcer, a Randomized Controlled Trial
Brief Title: Early Glue Saphenous Vein Ablation With Compression Versus Compression Alone in the Healing of the Venous Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI287/2560
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Venous Leg Ulcer
Keywords: Venous Leg Ulcer; Glue embolization; saphenous vein reflux
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: The randomised clinical trial with participants randomised1:1 to either:
  'Standard' therapy consisting of multilayer elastic compression bandaging/ stockings with deferred treatment of superficial reflux (usually once the ulcer has healed) Early endovenous glue embolization of superficial venous reflux(within 2 weeks) in addition to standard therapy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard therapy arm (Active Comparator): Multilayer elastic compression bandaging/ stockings with the deferred treatment of superficial reflux (usually once the ulcer has healed)
  Interventions: Procedure: Standard therapy arm
- Early endovenous glue embolization arm (Experimental): Early endovenous glue embolization of superficial venous reflux within 2 weeks in addition to standard compression therapy
  Interventions: Procedure: Early endovenous glue embolization arm

INTERVENTIONS:
Procedure: Standard therapy arm — Multilayer elastic compression bandaging/ stockings with the deferred treatment of superficial reflux (usually once the ulcer has healed)
  Arms: Standard therapy arm
Procedure: Early endovenous glue embolization arm — Early endovenous glue embolization of superficial venous reflux within 2 weeks in addition to standard compression therapy
  Arms: Early endovenous glue embolization arm

SUMMARY:
The study evaluates the effects of early endovenous glue ablation on ulcer healing in patients with chronic venous ulceration. Half the patients are randomized to receive early endovenous ablation (within 2 weeks) and a half to standard care

DETAILED DESCRIPTION:
To get the venous leg ulcer to heal, the current best treatment is to wear a multi-component compression bandage, with which about 60% of these ulcers will heal within 24 weeks. There is evidence that treatment of the varicose veins by surgery will prevent the ulcer from returning after it has healed. Recent studies have suggested that newer techniques of treating varicose veins, such as sclerotherapy, laser or radiofrequency in an outpatient setting may help the ulcers to heal more quickly and reduce the chance of the ulcer recurrence. The aim of this study is to see whether early treatment of varicose veins using endovenous glue embolization helps with healing.

ELIGIBILITY:
Inclusion Criteria:

* Current leg ulceration of greater than 6 weeks, but less than 6 months duration
* Able to give informed consent to participate in the study after reading the patient information documentation
* Patient age > 18 years
* Ankle Brachial Pressure Index (ABPI) ≥ 0.8
* Superficial venous disease on colour duplex assessment deemed to be significant enough to warrant ablation by the treating clinician (either primary or recurrent venous reflux)

Exclusion Criteria:

* Presence of deep venous occlusive disease or other conditions precluding superficial venous intervention
* Patients who are unable to tolerate any multilayer compression bandaging / stockings will be excluded.
* The inability of the patient to receive the prompt endovenous intervention
* Pregnancy (female participants of reproductive age will be eligible for inclusion in the study, subject to a negative pregnancy test prior to randomisation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to ulcer healing | time from date of randomisation to date of healing within the 12 month study period
  For the purposes of this study, ulcer healing is defined as complete re-epithelialization of all ulceration on the randomized (reference) leg in the absence of a scab (eschar) with no dressing required.

SECONDARY OUTCOMES:
Ulcer Healing Rate | 24 weeks & time to ulcer healing within the 12 month study period
  Healing rate will be reported at 24 weeks in addition to time to ulcer healing to allow comparison with other published studies
Ulcer recurrence / Ulcer Free Time | Up to 12 months
  Will be calculated up to 1 year for each study arm to allow a very practical and easily understood assessment of the clinical difference between the 2 arms of the study. This will also allow comparison with other studies that have reported this outcome. In order to facilitate accurate calculation of reoccurrence/ulcer free time, clinical follow up will be continued after ulcer healing up to 1 year after randomization.
Quality Of Life SF36 | 6 weeks post randomisation, 6 months, 12 months
  Generic (SF36) quality of life assessment
Quality Of Life CIVIQ-20 | 6 weeks post randomisation, 6 months, 12 months
  CIVIQ-20 assessment
Quality Of Life EQ5D | 6 weeks post randomisation, 6 months, 12 months
  Generic (EQ5D )quality of life assessment
Clinical Success - Presence of residual / recurrent varicose veins | at 6 weeks
  The presence of residual / recurrent varicose veins remaining on the venous duplex
Clinical Success - VCSS | at 6 weeks
  The Venous Clinical Severity Score (VCSS)
Clinical Success - Complications | up to 12 months
  Incidence of complications related to the endovenous intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nuttawut Sermsathanasawadi, MD, Principal Investigator — Mahidol University
Locations (1):
- Vascular Surgery, Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand